CLINICAL TRIAL: NCT06644326
Title: A Pharmacokinetic Bridging Study of Film-Coated Tablets of IkT-148009 in Older and Elderly Healthy Subjects
Brief Title: A PK Study of IkT-148009 in Older and Elderly Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ABLi Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: IkT-148009-103
Record Dates: First submitted 2024-09-12; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A IkT-148009 Dry/Wet (Active Comparator): 100mg IkT-148009 Wet & 100mg IkT-148009 Dry
  Interventions: Drug: 100mg IkT-148009 Wet; Drug: 100mg IkT-148009 Dry
- Part B - Ikt-148009 wet/ Itraconazole (Active Comparator): 200 mg Itraconazole & 50mg IkT-148009 Wet
  Interventions: Drug: 200 mg Itraconazole; Drug: 50mg IkT-148009 Wet

INTERVENTIONS:
Drug: 100mg IkT-148009 Wet — 100mg wet tablet formulation
  Arms: Part A IkT-148009 Dry/Wet
Drug: 200 mg Itraconazole — 2 100mg capsules
  Arms: Part B - Ikt-148009 wet/ Itraconazole
Drug: 100mg IkT-148009 Dry — 100mg dry tablet formulation
  Arms: Part A IkT-148009 Dry/Wet
Drug: 50mg IkT-148009 Wet — 50mg wet tablet formulation
  Arms: Part B - Ikt-148009 wet/ Itraconazole

SUMMARY:
This is a two-part study. Part A consists of two different IkT-148009-201 solid dosage formulations that are being evaluated to determine their steady-state pharmacokinetic profile.

Part B is a drug-drug interaction (DDI) study focused on evaluating the impact of a strong CYP3A inhibitor on the preferred dosage determined in part A.

DETAILED DESCRIPTION:
This is a two-part study.

Part A is a single dose (7-day) study to determine the safety, tolerability and pharmacokinetics (PK) of two different tablet formulations of IkT-148009 in older and elderly healthy subjects.

Subjects in each cohort of the study will be admitted to the unit the day prior to the expected day of dosing and will be confined to the unit for approximately 12 days. Each cohort will consist of six (6) subjects who will receive treatment with one of two formulations of IkT- 148009 film-coated tablets at a single dose once daily for 7 days.

Part B is a Drug-Drug Interaction (DDI) study to determine the effect of itraconazole on the pharmacokinetics of IkT-148009.

Subjects in each cohort of the study will be admitted to the unit the day prior to the expected day of dosing in each period and will be confined to the unit for approximately 6 days in period 1 and 10 days in period 2. Up to eight (8) subjects will be evaluated in a two-period design in the fed state.

In Period 1, the 50 mg film-coated IkT-148009 tablet dose pharmacokinetics will be measured, followed by a 7-day washout. In Period 2, the same eight subjects will first be administered a 200 mg once daily capsule dose of itraconazole for four days. On Period 2 day 4 subjects will take a single 200 mg capsule dose of itraconazole, followed one hour later by a 50 mg film-coated tablet dose of IkT-148009.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have all questions about the study answered and must have signed the informed consent document before any study-specific procedures are performed.
2. Healthy ambulatory male and female subjects with no history or evidence of clinically relevant medical disorders as determined by the Investigator in consultation with the Sponsor.
3. Bodyweight > 50 kg and body mass index (BMI) > 18.0 and < 32.0 kg/m2.
4. Physical examination, clinical laboratory values, vital signs, and electrocardiogram (ECG) data.
5. Female subjects must be postmenopausal, permanently sterile (bilateral tubal occlusion), or of childbearing potential with a negative pregnancy test, non-breastfeeding, and using two highly effective methods of birth control.
6. Male subjects must agree to practice an acceptable method of highly effective birth control.
7. Males must be willing to abstain from sperm donation from the screening visit, while on study and through 30 days after receiving the last dose of study drug.

Exclusion Criteria:

1. Any subject with previous exposure to imatinib or known hypersensitivity to imatinib.
2. Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at the screening and admission visits.
3. Clinically significant abnormal physical examination or 12-lead electrocardiogram (ECG) at the screening or admission visits.
4. Clinically significant abnormal renal function.
5. Significant history (within six months prior to receiving the study drug) and/or presence of hepatic, renal, cardiovascular, pulmonary, gastrointestinal, endocrinological, hematological, dermatological, psychiatric, neurological, immunologic, ophthalmologic, metabolic, fluid retention and edema, bleeding disorders including hemorrhage or oncological disease.
6. Any subject with a history, presence and/or current evidence of serologic positive result for hepatitis B surface antigen, hepatitis C antibodies, or HIV antibodies 1 or 2.
7. Recent history (within previous six months prior to screening) of alcohol or drug abuse (as judged by the investigator), or has consumed > 2 alcohol drinks/day during the last three months prior to screening.
8. Any subject who currently uses or has regularly used tobacco or tobacco-containing products (cigarettes, pipes, etc.) for at least 30 days prior to screening or positive urine cotinine screen at the screening or admission visits.
9. Any subject who has received treatment with an investigational drug during the 30 days prior to screening. Exposure to an investigational medical device within 30 days of screening.
10. Use of agents known to affect drug metabolism: use of any known CYP3A4 inducers and/or inhibitors or consumed grapefruit juice, grapefruit, Seville oranges or St John's Wort or products containing these within 14 days prior to first administration of study drug. Strong inducers of CYP3A4 include dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifampicin and phenobarbital. Strong inhibitors of CYP3A4 include ketoconazole, itroconazole, clarythromycin, atazanavir, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin and voriconazole.
11. Investigative site personnel or their immediate families (spouse, parent, child or sibling whether biological or legally adopted).
12. Any subject unwilling or unable to comply with study procedures.
13. Pregnant or nursing women.
14. Anyone who does not meet the requirements for exclusion of certain concomitant medications as defined in Section 7.5.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-08-17 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Patient Safety | Through study completion, an average of 17 days
  Changes in vital sign measurements including HR and blood pressure.
Patient Safety | Through study completion, an average of 17 days
  Changes in clinical laboratory data consisting of CBC, Serum Chemistry, FSH
Patient Safety | Through study completion, an average of 17 days
  Electrocardiogram [ECG] parameters of ventricular rate, RR or PR interval, QRS complex, and QTcF interval.
Patient Safety | Through study completion, an average of 17 days
  C-SSRS assessment values.
Pharmacokinetic parameters in the absence or presence of itraconazole: | Through study completion, an average of 17 days
  Pharmacokinetic parameters:
  • Area under the concentration-time curve from time zero to 96 hours (AUC0-∞)
Pharmacokinetic parameters in the absence or presence of itraconazole: | Through study completion, an average of 17 days
  Pharmacokinetic parameters:
  • Maximum plasma concentration (Cmax)
Pharmacokinetic parameters in the absence or presence of itraconazole: | Through study completion, an average of 17 days
  Pharmacokinetic parameters:
  • Area under the concentration-time curve from time zero to last time point (AUC0-last)
Assess the pharmacokinetics (PK) of IkT-148009 | Through study completion, an average of 17 days
  Pharmacokinetic parameters:
  • Area under the concentration-time curve from time zero to 96 hours (AUC0-∞)
Assess the pharmacokinetics (PK) of IkT-148009 | Through study completion, an average of 17 days
  Pharmacokinetic parameters:
  • Maximum plasma concentration (Cmax)
Assess the pharmacokinetics (PK) of IkT-148009 | Through study completion, an average of 17 days
  Pharmacokinetic parameters:
  • Area under the concentration-time curve from time zero to last time point (AUC0-last)
Patient Tolerability | Through study completion, an average of 17 days
  Adverse event reporting

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No